CLINICAL TRIAL: NCT04252352
Title: Treatment of Acne Scars With Fractional CO2 Laser Versus Radio-frequency Microneedling: A Randomized Controlled Trial
Brief Title: Treatment of Acne Scars With Fractional CO2 Laser Versus Radio-frequency Microneedling
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Aarhus University Hospital (Other)
Collaborators: Bispebjerg Hospital (Other)
Responsible Party: Sponsor
Organization: University of Aarhus (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CO2 laser vs radio-frequency
Record Dates: First submitted 2020-01-21; First posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Acne Scars - Mixed Atrophic and Hypertrophic
Keywords: Fractional CO2 laser; Radio-frequency microneedling
MeSH Terms: conditions — Hypertrophy

STUDY DESIGN:
Intervention Model Description: Intra-person split-face trial
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ablative fractional CO2 laser resurfacing (Active Comparator): One fractional CO2 laser treatment are performed of acne scars on one side of the face
  Interventions: Device: Ablative fractional CO2 laser resurfacing/Radio-frequency microneedling
- Radio-frequency microneedling (Active Comparator): One radio-frequency microneedling treatment are performed of acne scars on one side of the face
  Interventions: Device: Ablative fractional CO2 laser resurfacing/Radio-frequency microneedling

INTERVENTIONS:
Device: Ablative fractional CO2 laser resurfacing/Radio-frequency microneedling — Intra-person split-face trial
  Other Names: Fractional CO2 laser (Lumenis UltraPuls Encore laser system, Yokneam, Israel)/Radio-frequency microneedling device (LUTRONIC INFINI/ GENIUS, Goyang, Korea)

SUMMARY:
The study is a prospective, randomized, controlled, intra-person split-face trial with blinded evaluations. The objective is to compare efficacy and adverse effects of ablative fractional CO2 laser resurfacing versus radio-frequency microneedling for treatment of atrophic acne scars in the facial area. Two comparable areas with acne scars on each side of the face are treated. One area will be treated with fractional CO2 laser and the other area with radio-frequency microneedling.

Outcome measures will be assessed by blinded investigators and included subjects at baseline before treatment and at follow-up visits 2-4 days and 1 and 3 months post-treatment. On-site assessment and OCT will be performed at the time of the visits. OCT scans will be offered to the subjects and are optional. Clinical photos are used for documentation.

15 participants will be recruited. The participants will be recruited to enter the trial in the clinic by investigators at the Department of Dermatology, Bispebjerg Hospital, and must meet the inclusion criteria (at least 18 years of age, acne scars in the facial area, comparable atrophic acne scars on each side of the face, fitzpatrick skintype I-III) to be eligible to enter the study. No personal remuneration will be awarded the investigators. None of the collaborators have any personal economic interest in the study. Participants will not receive remuneration.

All treatments are performed at the Department of Bispebjerg Hospital and patients are covered by the Hospital's patient insurance.

The declaration of Helsinki will be respected as well as the standards of good clinical research. Respect for privacy as well as physically and mentally integrity of the participants will be maintained. The study will be performed in accordance with Danish Health care authorities.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Acne scars in the facial area (predominantly rolling scars)
* Comparable atrophic acne scars on each side of the face
* Fitzpatrick skintype I-III

Exclusion Criteria:

* Pregnant or nursing women
* Treatment with isotretinoin within the last 6 months
* Current treatment with NSAID and prednisolone
* Known tendencies to produce hypertrophic scars or keloids
* Infection in the treatment area
* Considered unable to follow the study protocol, e.g. alcohol dependence syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2020-02 (Estimated); Primary Completion 2020-10 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Asymmetry (scar texture, erythema, pigmentation) | 3 months
Patient satisfaction | 3 months
Adverse effects ( wounds, scars, pigmentation, erythema, edema) | 3 months
Optical coherence tomography | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: June Svendsen, Nurse, Study Director — Bispebjerg Hospital
Locations (1):
- Bispebjerg Hospital, Copenhagen, Copenhagen NV, Denmark

IPD SHARING:
Plan to Share IPD: No